CLINICAL TRIAL: NCT04329624
Title: The Effect of Perioperative LevosIMendan Administration on Postoperative N-terminal pRo Brain Natriuretic Peptide Concentration in Patients With Increased cardiOVascular Risk Factors Undergoing Noncardiac surgEry - A Double-blinded Randomized Clinical Trial
Brief Title: Effect Levosimendan Administration on Postoperative NT-proBNP in Cardiac Risk Patients
Acronym: IMPROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Edith Fleischmann, Ao. Univ. Prof. Dr. Edith Fleischmann, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPROVE_2.2
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Risk Factor
Keywords: Levosimendan; NT-proBNP; MINS; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan (Active Comparator): Patients receive a continuous infusion of 12.5mg solved in 50mL Levosimendan for up to 24 hours. Infusion will be started with surgical skin incision.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Patients receive a continuous infusion containing a placebo solved in 50mL for up to 24 hours. Infusion will be started with surgical skin incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Levosimendan 2.5 mg/ml injection contains levosimendan 2.5 mg, povidone 10.0 mg, citric acid, anhydrous 2.0 mg and ethanol, anhydrous to 1.0 mL. Levosimendan injection is a clear, yellow to orange solution. Immediately after skin incision patients allocated to the verum group will receive a dose of 12.5 mg in 500 mL of levosimendan.
  Arms: Levosimendan
Drug: Placebo — Placebo 2.5 mg/ml injection contains riboflavine sodium phosphate 0.4 mg, dehydrated alcohol 100 mg and water for injection to 1 mL.
  Immediately after skin incision patients allocated to the placebo group will receive 500 mL of 5% Glucose.
  Arms: Placebo

SUMMARY:
This is a prospective randomised trial investigating the effect of a preemptive administration of levosimendan on postoperative cardiac NT-proBNP concentrations.

DETAILED DESCRIPTION:
Major cardiovascular complications occur in about 3 % of all patients undergoing noncardiac surgery and are even higher in patients with increased preoperative risk factors. N-terminal pro brain natriuretic peptide (NT-proBNP) increases in over two third of patients undergoing surgery and is a strong predictor for perioperative myocardial complications. Levosimendan is a positive inotropic Ca2+ sensitizer and significantly reduces postoperative BNP concentration in cardiac surgery. The evidence in the non-cardiac surgery setting, however, is weak. Therefore, we will test our primary hypothesis that the perioperative administration of levosimendan significantly will reduce postoperative NT-proBNP concentrations in patients undergoing moderate- to high-risk non-cardiac surgery. We will also test the secondary hypotheses that levosimendan will reduce postoperative maximum troponin T (maxTnT) concentration, the incidence of myocardial injury after noncardiac surgery (MINS), myocardial infarction and death within 30 days and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

All patients need to meet all of the following criteria for inclusion (1-4):

1. Undergoing major surgery planned for more than 2 hours
2. ≥ 65 years of age and ≤ 85 years of age
3. Provide written informed consent AND
4. Fulfill ≥ 2 of the following criteria (A-E)

A) NT-proBNP ≥ 200 ng/L

B) History of coronary artery disease defined as 1 of the following 7 criteria (I to VII):

* I) History of angina
* II) History of myocardial infarction or acute coronary syndrome
* III) History of a segmental cardiac wall motion abnormality on echocardiography/radionuclide imaging
* IV) History of positive myocardial stress test (echocardiographic or radionuclide)
* V) History of a coronary artery stenosis > 50%
* VI) ECG with pathological Q waves in any two contiguous leads
* VII) History of previous artery revascularizations

C) History of permanent/paroxysmal atrial fibrillation diagnosed by physician/specialist

D) History of peripheral arterial disease as defined by a physician/specialist diagnosis of a current, or prior history of any 1 of the following 5criteria (I-V)

* I) Intermittent claudication
* II) Stenosis ≥ 70 % detected by angiography or doppler
* III) Stenosis ≤ 70% detected by angiography or doppler AND requiring medical treatment e.g. ASA or other platelet inhibitor
* IV) History of stroke or TIA - diagnosed by physician or CT/MRI
* V) Diagnosed cerebral arteriovascular disease (cAVK) diagnosed by a physician/specialist

E) Any 3 of 10 of the following risk criteria (i - x).

* i. History of congestive heart failure defined as a physician diagnosis of a current or prior episode of congestive heart failure OR prior radiographic evidence of vascular redistribution, interstitial pulmonary edema, or frank alveolar pulmonary edema;
* ii. History of a transient ischemic attack;
* iii. Diabetes and currently taking an oral hypoglycemic agent or insulin;
* iv. History of hypertension;
* v. Hyperlipidemia and currently taking a lipid lowering agent;
* vi. Documented chronic kidney disease diagnosed by physician/specialist and creatinine clearance > 30 ml/min
* vii. History of smoking within 2 years of surgery
* viii. Diastolic dysfunction (≥ grade 1) documented by echocardiography
* ix. Age ≥ 70 years
* x. Preoperative Troponin T (5th generation) ≥ 25ng/dL

Exclusion Criteria:

A) Previous adverse response and/or allergy to levosimendan B) ICU Patients undergoing surgery C) Preoperative Sepsis/SIRS needing ICU treatment D) Preoperative hemodynamically instable patients, who requirevasopressor or inotropic support E) Renal or liver transplantation F) History of severe heart failure (e.g. LVEF < 30%) G) Patients undergoing surgery for pheochromocytoma H) Liver cirrhosis I) Pulmonary hypertension (mPAP > 25 mmHg) J) Severe Renal Failure defines as creatinine clearance ≤ 30ml/min

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Postoperative maximum NT-proBNP concentration | First 5 Postoperative Days
  The administration of levosimendan improves LVEF and myocardial oxygen perfusion, which will be reflected in a decrease of postoperative NT-proBNP concentration.Since NT-proBNP is a strong predictor for postoperative cardiovascular complications in patients undergoing noncardiac surgery, we want to test the efficiency of levosimendan to decrease postoperative maxNT-proBNP concentrations in patients with increased cardiac risk factors undergoing moderate- to high-risk noncardiac surgery.

SECONDARY OUTCOMES:
Postoperative maximum troponin T concentration | First five postoperative days
  Levosimendan improves myocardial perfusion and might therefore reduce the postoperative maximum rise in TnT
Incidence of MINS (myocardial injury in non cardiac surgery) | First three postoperative days
  Levosimendan decreases the incidence of MINS during the first 3 postoperative days as compared to placebo in patients with increased cardiovascular risk factors undergoing moderateto high-risk noncardiac surgery. MINS is defined as: (i) a non-high-sensitivity troponin T >_30ng/L2 and (ii) a high-sensitivity troponin T (hsTnT) of 20 to <65 ng/L with an absolute change of at least 5 ng/L-this change threshold is independently associated with 30-day mortality [hazard ratio (HR) 4.69; 95% confidence interval (CI) 3.52-6.25]-or an hsTnT level >_65ng/ L. Furthermore, an absolute change of at least 5 ng/L is independently associated with 30-day mortality and will also be defined as MINS. TnT will be measured within 2 hours after surgery, on the first, second and third postoperative day.
Myocardial Infarction | 30 days and 1 year after surgery
  Levosimendan reduces the event rates of myocardial infarction and death during 30 days and 1 year after surgery as compared to placebo. Myocardial infarction is defined as a rise of TnT at least one value is above the 99th percentile URL and with at least one of the following: (i) symptoms of acute myocardial ischaemia; (ii) new ischaemic ECG changes; (iii) development of pathological Q waves; (iiii) imaging evidence of new loss of viable myocardium; (v) new regional wall motion abnormality in a pattern consistent with an ischemic ethiology; (vi) identification of a coronary thrombus by angiography including intracoronary imaging or autopsy.
Disability | 30 days and 1 year after surgery
  We evaluate the WHODAS 2.0 score before surgery on the day of consent, 30 days after surgery, and 1 year after surgery per phone call. For analyzing we use simply scoring. Each score is assigned to each of the following items - "none" (0), "mild" (1), "moderate" (2), "severe" (3), and "extreme (4).
  We will simply add up the scores from the items without recoding or collapsing of response categories, thus, there is no weighting of the individual items. As a result, the simple sum of the scores of the items across all domains constitutes a statistic that is sufficient to describe the degree of functional limitations.
NT-proBNP Mortality | 30 days and 1 year after surgery
  Perioperative NT-proBNP elevations are associated with postoperative mortality, cardiac mortality, mortality and nonfatal MI, and cardiac failure at both 30 days and 180 days or more after surgery.
  NT-proBNP values have been stratified to the previous published thresholds to predict mortality or MI after surgery.

OTHER OUTCOMES:
Sub-Study I: Fluid status determination | within 5 days after surgery
  Bioimpedance spectroscopy to determine perioperative fluid status including: 1) over hydration and total body water
Sub-Study II: Acute Kidney Injury | within 5 days after surgery
  The number of patients developing acute kidney injury after and the number of patients requiring renal replacement therapy after surgery.
Sub-Study III: Inflammatory Response | within 5 days after surgery
  Effect of levosimendan on postoperative maximum Interleukin 6 and CRP concentrations.
Sub-Study IV: Neurocognitive decline | within first 5 postoperative days and 1 year after surgery
  Effect of levosimendan on postoperative neurocognitive decline assess using MoCA

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodseth RN, Biccard BM, Chu R, Lurati Buse GA, Thabane L, Bakhai A, Bolliger D, Cagini L, Cahill TJ, Cardinale D, Chong CP, Cnotliwy M, Di Somma S, Fahrner R, Lim WK, Mahla E, Le Manach Y, Manikandan R, Pyun WB, Rajagopalan S, Radovic M, Schutt RC, Sessler DI, Suttie S, Vanniyasingam T, Waliszek M, Devereaux PJ. Postoperative B-type natriuretic peptide for prediction of major cardiac events in patients undergoing noncardiac surgery: systematic review and individual patient meta-analysis. Anesthesiology. 2013 Aug;119(2):270-83. doi: 10.1097/ALN.0b013e31829083f1. PMID 23528538
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Sessler DI, Meyhoff CS, Zimmerman NM, Mao G, Leslie K, Vasquez SM, Balaji P, Alvarez-Garcia J, Cavalcanti AB, Parlow JL, Rahate PV, Seeberger MD, Gossetti B, Walker SA, Premchand RK, Dahl RM, Duceppe E, Rodseth R, Botto F, Devereaux PJ. Period-dependent Associations between Hypotension during and for Four Days after Noncardiac Surgery and a Composite of Myocardial Infarction and Death: A Substudy of the POISE-2 Trial. Anesthesiology. 2018 Feb;128(2):317-327. doi: 10.1097/ALN.0000000000001985. PMID 29189290
- [Background] Rodseth RN, Biccard BM, Le Manach Y, Sessler DI, Lurati Buse GA, Thabane L, Schutt RC, Bolliger D, Cagini L, Cardinale D, Chong CP, Chu R, Cnotliwy M, Di Somma S, Fahrner R, Lim WK, Mahla E, Manikandan R, Puma F, Pyun WB, Radovic M, Rajagopalan S, Suttie S, Vanniyasingam T, van Gaal WJ, Waliszek M, Devereaux PJ. The prognostic value of pre-operative and post-operative B-type natriuretic peptides in patients undergoing noncardiac surgery: B-type natriuretic peptide and N-terminal fragment of pro-B-type natriuretic peptide: a systematic review and individual patient data meta-analysis. J Am Coll Cardiol. 2014 Jan 21;63(2):170-80. doi: 10.1016/j.jacc.2013.08.1630. Epub 2013 Sep 26. PMID 24076282
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Derived] Reiterer C, Kabon B, Taschner A, Graf A, Adamowitsch N, Horvath K, Emler D, Zotti O, Hantakova N, Hochreiter B, Fraunschiel M, Clement T, Fleischmann E. Levosimendan for postoperative subclinical heart failure after noncardiac surgery: a randomized, double-blinded, phase III trial. Nat Commun. 2025 Jul 1;16(1):5847. doi: 10.1038/s41467-025-60601-y. PMID 40593481
- [Derived] Reiterer C, Kabon B, Taschner A, Adamowitsch N, Graf A, Fraunschiel M, Horvath K, Kuhrn M, Clement T, Treskatsch S, Berger C, Fleischmann E. Effect of perioperative levosimendan administration on postoperative N-terminal pro-B-type natriuretic peptide concentration in patients with increased cardiovascular risk factors undergoing non-cardiac surgery: protocol for the double-blind, randomised, placebo-controlled IMPROVE trial. BMJ Open. 2022 Jan 21;12(1):e058216. doi: 10.1136/bmjopen-2021-058216. PMID 35063963